CLINICAL TRIAL: NCT06891534
Title: Circadian Regulation of Human Adipose Tissue Metabolism
Brief Title: Circadian Rhythms in Human Adipose
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Kelli A. Lytle, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 20-004280; K01DK140206 (NIH)
Record Dates: First submitted 2025-03-17; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-02

CONDITIONS: Obesity, Abdominal; Feeding Patterns
Keywords: circadian rhythms; adipose tissue; obesity; feeding pattern
MeSH Terms: conditions — Obesity, Abdominal; Feeding Behavior; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Normal weight participants (Active Comparator)
  Interventions: Other: Continuous Feeding; Other: Intermittent feeding
- Participants with obesity (Active Comparator)
  Interventions: Other: Continuous Feeding; Other: Intermittent feeding

INTERVENTIONS:
Other: Continuous Feeding — Participants will receive 24-hour continuous feeds through an NG tube
Other: Intermittent feeding — Participants will receive 3 boluses of feeding per day at regular meal times through an NG tube to mimic normal meals.

SUMMARY:
The goal of this study is to understand the underlying circadian rhythms in subcutaneous adipose tissue of humans with our without continuous feeding and how these are altered in people who have obesity.

DETAILED DESCRIPTION:
This proposal will address 3 main aims: 1) Determine the impact of endogenous AT circadian rhythms on AT function independent of diurnal nutrient delivery in humans, 2) determine the impact of central obesity on adipocyte circadian clock, and 3) establish for the first-time in vivo human adipocyte specific cistrome of the core circadian clock transcription factors, BMAL1 and CLOCK. In order to understand whether adipocytes have intrinsic circadian clock entrainment that is separate from food entrainment, we will compare rhythmicity of AT of lean volunteers studied under continuous vs. intermittent feeding paradigms. 20 normal weight adults (M/F= 10/10, split evenly between feeding groups) will be randomized to receive either "continuous" (CONT) feedings via a nasogastric (NG) feeding tube or receive 3 meals a day for the "intermittent" (INTER) study, also delivered via NG tube. The screening prior to the inpatient study visit will include vital signs, height, weight, hip/waist/neck circumference, body composition (DEXA scan) plasma lipid profile and fasting glucose. Potential volunteers will fill out questionnaires to exclude sleep disorders and assure normal sleep habits. For 3 days prior to and during the inpatient study, volunteers will be required to wear an Actiwatch 24 h/day; which objectively measures 24-hour sleep quality and quantity. (see detailed methodology).

For the inpatient visit, volunteers will be admitted to Mayo Clinic Clinical Research and Trials Unit (CRTU) at 1500 h where an NG tube will be placed. After baseline blood samples, the CONT feeding group will start liquid feedings (Ensure Plus®) at 1800 and continue for the next ~37 hrs. This will provide 12 h of continuous feeding before the first abdominal AT biopsies; this duration of continuous feeding abolishes the wide fluctuations in plasma insulin that occurs with normal meals and will avoid the progressive lipolytic response that would occur if fasting were used as the experimental design. FFA during isocaloric, continuous feeding is well within normal intraday variability. Participants randomized to INTER will receive 1/3rd of their daily energy needs at each "meal" via NG tube. These feedings will be given at 1800 h and 3 separate meals the following day. Participants will undergo measures of resting energy expenditure following the overnight period to appropriately interpret FFA Ra data.

To avoid retrieving AT sample from previously disrupted biopsy sites, every participant will be limited to 4 abdominal adipose tissue biopsies (1 per abdominal quadrant). To ensure a full 24 hours of data, all participants will have biopsies at: 0600, 1800, and 0600 the next day, half of participants will have a biopsy at 1200 and the other half at 2400. This hybrid (linked-cross sectional) will allow us to sample in series from multiple people and then create sample group means to account for disparate biopsy numbers. We are sampling from abdominal adipose tissue as this is the primary source of circulating FFA in humans and thus is the most likely for us to ascertain regulation of lipolysis proteins.

ELIGIBILITY:
Inclusion Criteria:

* BMI 20-25 kg/m2 or 30-37 kg/m2
* For participants with obesity a waist-to-hip ratio of ≥0.95 in males and ≥0.90 in females.
* sedentary
* females: non pregnant or breastfeeding
* ability to provide written informed consent and follow study instructions

Exclusion Criteria:

* History of mediations that impact adipocyte/lipid metabolism
* smoking
* insomnia
* sleep apnea
* sleep medication use
* employment in night or shift work
* extreme chronotypes
* Allergy to lidocaine

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-07-07 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
rhythmicity of circadian clock mRNA in adipose tissue | 24 hour
  Genes from RNA-seq analysis will be defined as statistically rhythmic.

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No